CLINICAL TRIAL: NCT01724164
Title: Robot- Versus Mirror-Assisted Motor Interventions in Rehabilitating Upper-Limb Motor and Muscle Performance and Daily Functions Poststroke: A Comparative Effectiveness Study
Brief Title: Robot- Versus Mirror-Assisted Rehabilitation in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201003058R
Record Dates: First submitted 2012-08-28; First posted 2012-11-09 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy; proto-oncogene protein c-fes-fps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Robotic assisted therapy (Experimental): This protocol includes 5 to 10 min of warm-up, 1 hr of RR, and 15 to 20 min of functional activities training. The treatment intensity is 1.5 hours/day, 5days/week for 4 consecutive weeks. The RR session uses the robot-assisted arm trainer, Bi-Manu-Track (Reha-Stim Co., Berlin, Germany).
  Interventions: Behavioral: Robotic assisted therapy
- Mirror Therapy (Experimental): This protocol includes 1 hour mirror therapy and 0.5 hour functional training in a session. The treatment intensity is 1.5 hours/day, 5 days/week, for 4 weeks. MT focuses on symmetrical bimanual movements and simultaneously observing the mirror visual feedback reflected by the unaffected upper extremity.
  Interventions: Behavioral: Mirror Therapy
- Conventional Rehabilitation (Active Comparator): Participants in this group receive a structured protocol based on occupational therapy such as neuro-developmental techniques and task-oriented approach. The treatment dose is matched to RR and MT groups.
  Interventions: Behavioral: Conventional Rehabilitation
- Robotic rehabilitation with FES (Experimental): This combined RR-FES treatment involves the same protocol as the RR regimen except that patients receive FES concurrently with RR.
  Interventions: Behavioral: Robotic rehabilitation with FES
- Robotic Rehabilitation with PI (Placebo Comparator): The RR-PI protocol is the same as the RR-FES protocol described above except that the surface electrodes are attached to the same target muscles on the affected upper limb but there is no output of electrical stimulation.
  Interventions: Behavioral: Robotic Rehabilitation with PI

INTERVENTIONS:
Behavioral: Mirror Therapy — This protocol includes 1 hour mirror therapy and 0.5 hour functional training in a session. The treatment intensity is 1.5 hours/day, 5 days/week, for 4 weeks. MT focuses on symmetrical bimanual movements and simultaneously observing the mirror visual feedback reflected by the unaffected upper extremity.
  Other Names: MT
  Arms: Mirror Therapy
Behavioral: Robotic assisted therapy — This protocol includes 5 to 10 min of warm-up, 1 hr of RR, and 15 to 20 min of functional activities training. The treatment intensity is 1.5 hours/day, 5days/week for 4 consecutive weeks. The RR session uses the robot-assisted arm trainer, Bi-Manu-Track (Reha-Stim Co., Berlin, Germany).
  Other Names: RT
  Arms: Robotic assisted therapy
Behavioral: Robotic Rehabilitation with PI — The RR-PI protocol is the same as the RR-FES protocol described above except that the surface electrodes are attached to the same target muscles on the affected upper limb but there is no output of electrical stimulation.
  Other Names: RR with Placebo Intervention (RR-PI)
  Arms: Robotic Rehabilitation with PI
Behavioral: Robotic rehabilitation with FES — This combined RR-FES treatment involves the same protocol as the RR regimen except that patients receive FES concurrently with RR.
  Other Names: RR combined Functional Electrical Stimulation (RR-FES)
  Arms: Robotic rehabilitation with FES
Behavioral: Conventional Rehabilitation — Participants in this group receive a structured protocol based on occupational therapy such as neuro-developmental techniques and task-oriented approach. The treatment dose is matched to RR and MT groups.
  Other Names: CR; Control Treatment; CT
  Arms: Conventional Rehabilitation

SUMMARY:
The purpose of this proposal is 1) to compare the relative effects of the robotic rehabilitation (RR), mirror therapy (MT), and conventional intervention (CI), 2) to compare the effects of the combined therapy of the RR-Functional Electrical Stimulation (FES) and the RR-Placebo Intervention (PI), and 3) to identify the clinical predictors that will potentially influence the functional outcomes after interventions.

DETAILED DESCRIPTION:
Emerging stroke rehabilitation therapies have shown promise for improving motor recovery after stroke and involve elements of high-intensity and repetitive task-specific practice, which might be the essential elements of treatment success. Two prominent examples of advances in innovative rehabilitation therapies after stroke include robotic rehabilitation (RR) and mirror therapy (MT). Based on the development of mechanical and biomedical engineering, RR has emerged that incorporates therapeutic elements for success in motor rehabilitation: high-intensity, repetitiveness, task-specificity, feedback, and bilateral training into its design. MT has been proposed in the light of translational research of mirror neurons. In MT, patients place a mirror beside the unaffected limb to block their view of the affected limb, creating the illusion that both limbs are intact. The motor visual input from MT facilitates the activations in the premotor, primary motor and somatosensory areas, which enhance sensory, perception and motor abilities. The MT may be used to restore sensory functions, improve grip/grasp strength and motor function. In addition, an innovative technology, functional electrical stimulation (FES), is proposed as an adjunct to assist in movement execution and increase the electric activity of muscles for movement and the active range of motion in patients with low functioning. Robotic rehabilitation that emphasizes muscle strengthening and motor restoration may be implemented in combination with the FES to improve treatment outcomes in stroke patients with moderate-to-severe motor impairments in movement performance and functional outcomes. Despite these promises, research studies that investigate comparative efficacy of the rival therapies and the effects of combined therapy relative to mono-therapy are lacking. An additional gap in contemporary neurorehabilitation is the lack of sufficient information on the threshold values of clinically significant change in a variety of functional domains relevant for individualized medicine. In addition, research on the potential vales of biomarkers (eg, level of oxidative stress) for use in outcomes study in intense rehabilitation falls far behind disciplines of basic sciences. This proposed research project will be devoted to comparative efficacy trials and clinimetric study to promote evidence-based neurorehabilitation and translational research in stroke.

It has been called for comparative effectiveness research of the innovative treatments to promote evidence-based practice and translational science in stroke motor rehabilitation. Scientific evidence for comparative effectiveness research of RR versus MT on functional outcomes (e.g., motor, muscle, sensory, and daily functions) and adverse physiological responses (e.g., fatigue and oxidative responses) in stroke patients is limited. More rigorous studies are needed to compare the efficacy of RR and MT with control intervention (CI), to identify the predictors of treatment success, and to study change in functions (motor, muscle, sensory, and daily) and level of fatigue and oxidative stress after intense training in order to promote translational science in movement therapy. Therefore, this comparative efficacy research aims at performing a randomized controlled trial (RCT) to (1) verify the efficacy and motor control mechanisms of dose-matched RR, MT, and CI; (2) examine whether RR combined with FES will enhance the effect of RR; (3) study the predictors of treatment outcomes and clinimetric properties of the outcome measures. We hypothesize the RR and MT groups would produce better performance in motor control, muscle function, sensory function, daily functions, and quality of life than the CI group. We further hypothesize that there will be a differential improvements in movement performance and sensory functions between the RR and MT. Combined therapy of the RR and FES (RR-FES) will enhance the effect of RR as compared with the RR plus placebo intervention (RR-PI).

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide the written informed consent
* More than 6 months onset of unilateral stroke
* An initial 25-56 or 18-50 scores on the upper limb subtest of the Fugl-Meyer assessment (FMA)
* Sufficient cognitive ability (Mini Mental State Examination ≧ 24 points)
* Without upper limb fracture within 3 months

Exclusion Criteria:

* Recurrent of stroke or seizure episode during the intervention
* Occurrence of serious or continuous pain on affected upper-extremity
* History of other neurological disease or severe orthopaedic condition

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-01 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | 2011/8 to 2013/1 (up to 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Keh-chung Lin, ScD, Principal Investigator — School of Occupational Therapy, College of Medicine, National Taiwan University
Locations (2):
- Taiwan (2):
  - National Taiwan University Hosipital, Taipei, Taiwan
  - National Taiwan University Hospital, Taipei, Taiwan